CLINICAL TRIAL: NCT03582579
Title: Enhancing Brain Training With Virtual Reality
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: NeuroTrainer (Industry)
Responsible Party: Principal Investigator, Duje Tadin, Associate Professor, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 70869
Record Dates: First submitted 2018-03-20; First posted 2018-07-11 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control in VR (Experimental): Adults ages 18 to 35 who will be training in Virtual Reality.
  Interventions: Behavioral: Training in Virtual Reality
- Control Non-VR (Experimental): Adults ages 18 to 35 who will be training on a computer screen.
  Interventions: Behavioral: Training on a computer screen
- College Athletes with TBI Group (Experimental): Adults ages 18 to 35 with mild TBI who will be training in Virtual Reality
  Interventions: Behavioral: Training in Virtual Reality
- Older Adult Group (Experimental): Older Adults over the age of 65 who will be training in Virtual Reality
  Interventions: Behavioral: Training in Virtual Reality

INTERVENTIONS:
Behavioral: Training in Virtual Reality — Action Video Game Based Training in Virtual Reality
  Arms: College Athletes with TBI Group; Control in VR; Older Adult Group
Behavioral: Training on a computer screen — Action Video Game Based Training on a computer screen
  Arms: Control Non-VR

SUMMARY:
The purpose of this study is to evaluate the effectiveness of brain training in a Virtual Reality set up in neurotypical populations as well as in the traumatic brain injury population.

DETAILED DESCRIPTION:
Brain training is a large and a growing field, both scientifically and commercially. Emerging evidence demonstrates that training can promote beneficial brain plasticity in both healthy individuals and clinical populations. Much of the recent interest in brain training can be traced back to the seminal work done at the University of Rochester, where Daphne Bavelier and colleagues showed that training with action video games (AVG) can lead to a wide range of cognitive and perceptual improvements. In our recent work, we developed a novel training paradigm that isolates and concentrates the key aspects of AVG-training while eliminating complex and often violent gameplay associated with AVGs. The results revealed similarly broad effects of training as with conventional AVGs. In this study, we aim to move this training paradigm to virtual reality (VR) and extend its application to cognitive aging and mild traumatic brain injury (TBI) populations.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is an adult over the age of 18.
* Has the capacity to give consent.
* Has normal or corrected to normal vision.
* Has adequate hearing.
* Is a non-action video game player.
* Is a non-VR game player. All subjects will be assigned to one of four groups: a Control Group training in VR, a Control Groups training on a 2D display, an Older Adult Group without dementia training in VR, and a College Athletes with mild TBI Group training in VR.

Specific Inclusion Criteria for both Control Groups. The subject must:

* Be between the ages of 18 and 35.
* Have no neurologic or vascular disorders/injuries.

Specific Inclusion Criteria for the College Athletes with TBI Group. The subject must:

* Be between the ages of 18 and 35.
* Be diagnosed with mild TBI (i.e., concussion) within the last two weeks.

Specific Inclusion Criteria for the Older Adult Group. The subject must:

* Be over the age of 65.
* Have no neurologic or vascular disorders/injuries.

Exclusion Criteria:

A person will be excluded from the study if he/she:

• Is under the age of 18.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-06-27 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Visual Crowding (a measure of spacial resolution of attention) | 6 weeks
  This is a visual task which will be done an a computer twice. Once prior to the start of training and then again following training. The results (including the number of trials correct as well as the time it took for the subject to respond) will be analyzed and compared across groups.
Attentional Blink (a measure of temporal resolution of attention) | 6 weeks
  This is a visual task which will be done an a computer twice. Once prior to the start of training and then again following training. The results (including the number of trials correct as well as the time it took for the subject to respond) will be analyzed and compared across groups.
Useful Field of View (a measure of spacial awareness) | 6 weeks
  This is a visual task which will be done an a computer twice. Once prior to the start of training and then again following training. The results (including the number of trials correct as well as the time it took for the subject to respond) will be analyzed and compared across groups.

CONTACTS AND LOCATIONS:
Overall Officials: Duje Tadin, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided